CLINICAL TRIAL: NCT03327766
Title: Assesment of Vit D3 Level in Cases of Unexplaind Pregnancy Loss in Assiut
Acronym: vitDinRPL
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Woman's Health University Hospital, Egypt (Other)
Responsible Party: Principal Investigator, Hisham Ahmed El-Sayed Abou-Taleb, lecturer of obstetrics and gynecology, Woman's Health University Hospital, Egypt
Other Study IDs: Vit D and RPL
Record Dates: First submitted 2017-10-27; First posted 2017-10-31 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: vitD3 Level in Cases of Recuurent Pregnancy Loss
Keywords: vitamin D and recurrent pregnancy loss

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum samples from both cases and control groups will be stored at -20 degrees
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RPL group: history of unexplained recurrent pregnancy loss (defined as two or more consecutive missed miscarriage before 14 weeks of gestation).
  Interventions: Diagnostic Test: 4-Measurment of serum 25(OH)D3 using Vidas by ELFA meathod.
- Control group: womens coming for contraception after normal pregnancy outcome.
  Interventions: Diagnostic Test: 4-Measurment of serum 25(OH)D3 using Vidas by ELFA meathod.

INTERVENTIONS:
Diagnostic Test: 4-Measurment of serum 25(OH)D3 using Vidas by ELFA meathod. — A specialized test of the 25(OH)D serum level was conducted and the blood samples were collected in the months of November to April. The winter months were chosen intentionally in order to limit the impact of the sun light upon 25(OH)D serum level.The test VIDAS® 25 OH Vitamin D Total was used-enzyme immunoassay with highly fluorescent measurement ELFA. According to the reference values of this method the 25(OH)D < 20 ng/ml serum levels are considered as deficiency and the serum levels between 20 - 30ng/ml are defined as insufficiency. It's sufficient if the level of 25(OH)D is 30 to 100 ng/ml.

SUMMARY:
Assesment of Vit D3 leve in cases of unexplained recurrent pregnancy loss in assiut

DETAILED DESCRIPTION:
Recurrent pregnancy loss is defined as two or more consecutive pregnancy loss before 20 weekse of gestation (1). It affects about 1-5% of women of reproductive age. This not only causes significant physical and mental problems in families, but also a heavy economic burden on families and health systems (2, 3) Recurrent pregnancy loss (RPL) is a syndrome caused by multiple etiologies such as anatomical, endocrine, genetic, infectious, immunological, thrombotic and unexplained etiologies hence an investigation of underlying etiologies is often complicated When the conventional investigation scheme is applied, up to 60% of women with RPL remain unexplained (4). Recent studies have indicated that immune inflammatory and thrombotic conditions are two major under-lying pathologies for RPL (5). Approximately 20% of women with RPL have autoimmune conditions, such as antiphospholipid antibody (APA)(6),antinuclear antibody (ANA), anti-thyroperoxidase antibody and anti-thyroglobulin antibody(7,8).

Immune function in pregnancy From initial implantation of the conceptus, the maternal uterine endometrium undergoes decidualisation to support placental development and function. The resulting decidua is a tissue formed from the maternal endometrium, originating from epithelial and stromal cells, and is characterised by invasion from the extraembryonic fetal-derived trophoblasts and close 'cell-cell juxtaposition' of these different tissues The principal function of the decidua is to facilitate early fetal-maternal exchange of nutrients, gases and waste, while also acting as a secretory source of steroid hormones, cytokines and growth factors (9).However, the decidua also plays a key role in protecting pregnancy against maternal immune surveillance(10) .

Cellular infiltration is a key feature of immune function within decidua, and leukocytes comprise at least 40% of the total decidual stromal cell population(11) . The leukocyte subtypes present include decidual (uterine) natural killer (uNK) cells, macrophage subtypes, CD4C and CD8C T-lymphocytes (including T-regulatory cells (Tregs) and antigen-presenting cells (APCs) such as dendritic cells (DCs)(12) . There has been renewed interest in the role vitamin D, as key regulators of decidual immune cell function and its roles in fetal-maternal immune tolerance (13) .

- 3 - Vitamin D and autoimmunity Vitamin D, a steroid hormone, is well known to be involved in calcium and phosphate homeostasis and bone metabolism (14).The target organs for the non-classical actions of the vitamin D include immune systems, pancreatic b-cells, the heart and cardiovascular system, the brain and reproductive tissues. Tissue responses to vitamin D include regulation of hormone secretion modulation of immune responses, and a control of cellular proliferation and differentiation (15). Vitamin D was also reported to inhibit proliferation of T helper 1 (Th1) cells and limit their production of cytokines, such as interferon gamma (IFN-g), interleukin-2 (IL-2) and tumor necrosis factor-alpha (TNF-a).Conversely, vitamin D induces T helper 2 (Th2) cytokines, such as IL-4, IL-5, IL-6, IL-9, IL-10 and IL-13 (16). Furthermore, in many studies vitamin D has been presented as a modifiable environmental factor for Th1-mediated autoimmune disease and appears to be important for susceptibility to and severity of the disease (17). Vitamin D also regulates B cell immunity. It down-regulates the proliferation and differentiation of B lymphocytes and inhibits IgG production (16).

Vitamin D deficiency in pregnant women is associated with increased risk of obstetrical complications such as pre-eclampsia (18), bacterial vaginosis associated preterm delivery (19), gestational diabetes mellitus (20) and small-for-gestational age births (21).

ELIGIBILITY:
Inclusion Criteria:

1. Age of women 20:35years old
2. history of unexplained recurrent pregnancy loss (defined as two or more consecutive missed miscarriage before 14 weeks of gestation).

Exclusion Criteria:

1. Un corrected uterine anomalies.
2. Uncontrolled DM .
3. Systemic disease(SLE,Rheumatoid arthritis).
4. Thyroid dysfunction.
5. Antiphospholipid antibody syndrome
6. Cervical incompetence

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 50 womens with history of RPL in last 2 pregnanses and last abortion of 6 months at El-mabra H. & AUH.
  50 womens coming for contraception after normal pregnancy outcome. As acotrol group.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2018-04-30 (Estimated); Study Completion 2018-10-31 (Estimated)

PRIMARY OUTCOMES:
vitamin D level | 1 year
  the serum level of will be checked in ng/ml

CONTACTS AND LOCATIONS:
Overall Officials: Ezat Hamed, Study Director — Professor of obstetrics and gynecology Faculty of medicine-Assiut university

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hou W, Yan XT, Bai CM, Zhang XW, Hui LY, Yu XW. Decreased serum vitamin D levels in early spontaneous pregnancy loss. Eur J Clin Nutr. 2016 Sep;70(9):1004-8. doi: 10.1038/ejcn.2016.83. Epub 2016 May 25. PMID 27222154